CLINICAL TRIAL: NCT02488837
Title: Investigation of Non-Invasive Outcomes Predictors in Patients Undergoing Deep Brain Stimulation for Movement Disorders
Brief Title: Investigation of Non-Invasive Outcomes Predictors in Patients Undergoing DBS for Movement Disorders
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Harrison Walker, MD, Associate Professor of Neurology, University of Alabama at Birmingham
Other Study IDs: F140225003
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Movement Disorders
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DBS subjects: deep brain stimulation (DBS) in patients with Parkinson's disease, tremor, dystonia, and Tourette's syndrome

SUMMARY:
The purpose of the study is to determine if non-invasive measurements of brain waves from the skin called electroencephalography (EEG) can predict whether the brain stimulator will help your symptoms. Our goal is to obtain these brain wave measurements with patients both awake and under general anesthesia, and then to evaluate which brain wave patterns are associated with clinical improvement to determine if they could be useful for predicting whether the surgery will work. If such predictive measures were established based upon the findings of this study, they could be used in the future to improve surgical outcomes in the following ways: (1) to help guide surgical targeting in the operating room awake or under anesthesia, (2) to guide post-operative programming in clinic, and (3) and to develop potential feedback systems for "automatic" programming of the brain stimulator system at home.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who elect to undergo deep brain stimulation as part of routine clinical care for movement disorders (Parkinson's disease, essential tremor, dystonia, Tourette's syndrome).
2. Adults, ages 19 and older

Exclusion Criteria:

1. Patients who are outside the age range for inclusion
2. Patients who are unable to consent to the research for cognitive or behavioral reasons
3. Patients who are medically too ill to participate, and
4. Patients who have their DBS programming at outside facilities

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo deep brain stimulation as part of routine clinical care for movement disorders (Parkinson's disease, essential tremor, dystonia, Tourette's syndrome).
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Change in the rating scale score at 6 months post-op versus pre-op baseline
  Validated rating scale for measuring symptoms of Parkinson's disease
The Essential Tremor Rating Assessment Scale (TETRAS) | Change in the rating scale score at 6 months post-op versus pre-op baseline
  Validated rating scale for measuring symptoms of essential tremor
Burke-Fahn-Marsden (BFM) Dystonia Rating Scale | Change in the rating scale score at 6 months post-op versus pre-op baseline
  Validated rating scale for measuring symptoms of primary dystonia
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | Change in the rating scale score at 6 months post-op versus pre-op baseline
  Validated rating scale for measuring symptoms of primary cervical/segmental dystonia
Yale Global Tic Severity Scale | Change in the rating scale score at 6 months post-op versus pre-op baseline
  Validated rating scale for tic severity
Deep Brain Stimulation (DBS) Therapeutic Window | 1 month post-operative scores for each contact on the DBS electrode array
  Measurement of the available range of stimulation intensities for therapy for each contact on the DBS electrode array

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Walker, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States